CLINICAL TRIAL: NCT06354517
Title: The Impact of the SENSE Program on Parent and Newborn
Brief Title: The Impact of the SENSE Program on NICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Mujde CALIKUSU INCEKAR, Associate Professor, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YIU-M-CI-003
Record Dates: First submitted 2024-03-29; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pre-Term; Individualized Developmental Care; Sensory Experiences
MeSH Terms: conditions — Premature Birth | interventions — Social Cohesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SENSE group (Experimental): Parents of babies in this group will be given SENSE program training. After the training, parents will care for their babies within the scope of the SENSE program. These babies will receive care from their parents with positive sensory exposures within the scope of the SENSE program from admission to the clinic until discharge. Data collection forms will be administered to babies and their parents.
  Interventions: Other: SENSE group
- Control group (No Intervention): The SENSE program will not be applied to the parents of babies in this group. These babies will receive the routine care of the clinic. These babies will be monitored from admission to the clinic until discharge. Data collection forms will be administered to infants and parents.

INTERVENTIONS:
Other: SENSE group — Parents of babies in this group will be given SENSE program training. After the training, parents will care for their babies within the scope of the SENSE program. These babies will receive care from their parents with positive sensory exposures within the scope of the SENSE program from admission to the clinic until discharge. Data collection forms will be administered to babies and their parents.
  Arms: SENSE group

SUMMARY:
The SENSE program will be applied to babies receiving treatment in the neonatal intensive care unit and the effect of the application on the baby and parents will be examined.

DETAILED DESCRIPTION:
For the growth and health of the baby, the intrauterine environment provides the fetus with protective physical barriers and sensory exposures timed appropriately for its development. These early exposures occur during sensory development in the intrauterine environment, and there are differences in the timing of development of each sense. When the baby is born prematurely, the intrauterine environment is replaced by the Neonatal Intensive Care Unit environment. The sensory environment of the preterm baby includes the experiences of touch, movement, smell, sound, light, frequent nociceptive pain and disruption of sleep. The mismatch between the infant's underdeveloped coping skills and the stimulating NICU environment can cause physiological imbalance, negatively impact growth and development, and ultimately predispose to the development of long-term neurodevelopmental consequences. Although harmful sensory exposures can negatively affect the development of the preterm baby, appropriate positive sensory exposures positively affect brain development.

ELIGIBILITY:
Inclusion Criteria:

* Being in the first week of life

Exclusion Criteria:

* Congenital anomaly,
* Preterm babies who are not predicted to survive,
* Babies who cannot be followed regularly,
* Parent having a psychiatric problem
* Parents who wish to withdraw from the study

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Hammersmıth Neonatal Neurologıcal Examınatıon | 24 hours
  It will be applied twice: when the baby is first admitted to the clinic and before discharge.
Parental Stress Scale: Neonatal Intensive Care Unit | 24 hours
  It will be applied twice: when the baby is first admitted to the clinic and before discharge.
State-trait Anxiety Inventory | 24 hours
  It will be applied twice: when the baby is first admitted to the clinic and before discharge.
Edinburgh Postnatal Depression Scale | 24 hours
  It will be applied twice: when the baby is first admitted to the clinic and before discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim SAVAŞER, PhD, Principal Investigator — Biruni University; Ahu ÇIRLAK, PhD, Principal Investigator — Ankara Guven Hospital
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)